CLINICAL TRIAL: NCT02120144
Title: Effect of Observation Plus Imagination of Gait on Stride Variability in Young and Older Adults
Acronym: OBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-A00829-36
Record Dates: First submitted 2014-03-12; First posted 2014-04-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2014-03

CONDITIONS: Gait Variability; Elders; Fall; Re-education
MeSH Terms: interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 15 young patients (<65 years old) and 15 older patients (>64 years old) are submitted to an observation phase and an imagination phase of walking at a precise rythm for 10 minutes
  Interventions: Other: Observation & imagination
- Reading (Active Comparator): 15 young patients (<65 years old) and 15 older patients (>64 years old) are submitted to a reading phase on a computer for 10 minutes.
  Interventions: Other: Reading

INTERVENTIONS:
Other: Observation & imagination — It is a combination of an observation phase followed by an immediate imagination phase of a straight gait with an imposed cadency.
  Arms: Intervention
Other: Reading — A 10 minutes reading phase of François Mauriac's "Therese Desqueyroux" on a computer
  Arms: Reading

SUMMARY:
The aim of study is to examine the combined effect of observation and imagination of gait on stride time variability of stride time among in healthy young and older adults.

DETAILED DESCRIPTION:
JUSTIFICATION :

* In geriatric rehabilitation, gait reeducation, especially after a fall, is often encountered at the very beginning, to the inability to walk again. The main reasons are poorly controlled pain, immobilisations of a segment or the entire lower limb and adaptation to certain prostheses after fracture. This delay in walking recovery leads briefly to acute postural disadaptation that exposes to multiple decubitus complications such as infections, bedsores and muscular atrophy. Conventional rehabilitation techniques are then difficult to implement because they are poorly adapted to the geriatric patients.
* Today, many experimental data suggest a functional equivalence between making a movement, imagining and observing it. These data can be used to support the development of new rehabilitation techniques. For example, mental imagery is used in the learning of complex movements in order to improve motor performance.
* Stride variability, and more specifically stride time variability was identified as the best marker of the automatic walking, a low variability corresponding to an automatic and safety gait.
* We hypothesize that the combined effect of observation and imagination of a gait using an imposed cadency cadency may reduce stride time variability of stride time in healthy young and older adults.

The secondary objectives of the study are as follows:

* To examine the combined effect of observation and imagination of a gait on mean value of spatio-temporal parameters in healthy young and older adults.
* To study the influence of age on the combined effect of observation and imagination of gait on mean value and coefficient of variation of spatio-temporal parameters in healthy young and older adults

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Able to walk without walking aid on 15 metres
* Written informed consent to participate in the study (or trustworthy person)
* Being affiliated to a social security regime

Exclusion Criteria:

* Osteoarticular pathologies of the lower limbs and / or spine altering the biomechanical characteristics of the body members.
* Ataxia
* History and / or progressive neuropsychiatric disorders.
* Score in the 4-items Geriatric Depression Scale > 1.
* Enrolment in another simultaneous clinical trial (Participation in a concomitant clinical trial.)
* Civil defense measures underway (Measures civil protection type trusteeship / guardianship / safeguarding justice in progress.)
* Refusal to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mean value of stride time variability | this outcome is assessed at baseline and 10 minutes later.
  measured by the coefficient of variation (COV= standard deviation/Average) x 100.

SECONDARY OUTCOMES:
Average value of all spatio-temporal gait parameters and age. | this outcome is assessed at baseline and 10 minutes later.
Clinical characteristics of participants | this outcome is assessed at baseline.
  Age. Gender. Medical and surgical history. Age of acquisition of walking Practice of regular physical activity. Practice of sport. Personal characteristics: weight, size, height of the lower limbs. Number of different therapeutic classes taken per day. Proprioception of lower limb using a graduated diapason (normal maximum score of 8)

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, Maine et Loire, France